CLINICAL TRIAL: NCT04899557
Title: Retrospective/Prospective Study of Pediatric Surgical Patients
Status: Completed | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Greg Klazura, Pediatric Global Surgery Fellow, University of Illinois at Chicago
Other Study IDs: 2014-0396
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2021-05

CONDITIONS: Pediatric Robotic Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Procedure: Single Port Robotic Splenectomy — Pediatric patient with splenomegaly underwent a single port robotic splenectomy.

SUMMARY:
UIC Division of pediatric surgery has IRB approval to perform retrospective and prospective study of their pediatric surgical patients. At UIC Dr. Lobe performed the first known single port robotic splenectomy on a child and as a surgical first this case is worthy of a case report. Since it is a surgical and therapeutic first it needs to be aon regestiry of health research prior to publication.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patient with splenomegaly

Exclusion Criteria:

* NOn pediatric patients

Ages: 0 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: pediatric patient with splenomegaly
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days post op
  Did the patient die from the operation

CONTACTS AND LOCATIONS:
Overall Officials: Greg Klazura, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Office for the Protection of Research Subjects, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No